CLINICAL TRIAL: NCT03071536
Title: Furosemide Stress Test as a Marker of Postoperative Kidney Allograft Function
Brief Title: Furosemide Stress Test Predicting Early Graft Function in Kidney Transplantation
Acronym: FOSTIK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Suwasin Udomkarnjananun, Suwasin Udomkarnjananun, M.D., King Chulalongkorn Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 317/59
Record Dates: First submitted 2017-02-20; First posted 2017-03-07 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Kidney Function; Kidney Transplant; Complications; Delayed Graft Function
Keywords: furosemide stress test; kidney transplantation; urine output; perioperation; delayed graft function
MeSH Terms: conditions — Delayed Graft Function | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furosemide (Experimental): Single dose of furosemide 1.5 mg/kg intravenously will be given to all participants at 3 hours post-reperfusion of kidney allograft.
  Urine output will be recorded hourly for 6 hours.
  Interventions: Drug: Furosemide Injection

INTERVENTIONS:
Drug: Furosemide Injection — Furosemide 1.5 mg/kg intravenously at 3 hours post-reperfusion of kidney allograft

SUMMARY:
Furosemide is an old drug that has been used frequently in the postoperative period of kidney transplantation, aiming to achieve adequate urine output. There is no previous study that directly evaluate the urine response to standardized dose of furosemide in the postoperative period. The objective is to measure the urine output after standardized dose of furosemide is delivered, as a biomarker to predict the graft function in perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Deceased donor kidney transplantation at KCMH
* informed consent is accepted

Exclusion Criteria:

* Known allergy to furosemide
* Surgical complication of allograft
* Urgently needed for dialysis (refractory hypervolemia, uremic symptoms, and hyperkalemia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-11-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Urine output | 6 hours
  Urine output per hour (milliliters/hour) after furosemide injection

SECONDARY OUTCOMES:
Delayed graft function | 7 days
  Delayed graft function is defined by the necessity of dialysis within the first week after kidney transplantation. (yes/no)
Creatinine reduction ratio | At postoperative day 0,7 and 14
  Ratio of serum creatinine at postoperative day 7 and 14 to day-zero creatinine

CONTACTS AND LOCATIONS:
Overall Officials: suwasin udomkarnjananun, M.D., Principal Investigator — King Chulalongkorn Memorial Hospital and Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Udomkarnjananun S, Townamchai N, Iampenkhae K, Petchlorlian A, Srisawat N, Katavetin P, Sutherasan M, Santingamkun A, Praditpornsilpa K, Eiam-Ong S, Avihingsanon Y. Furosemide Stress Test as a Predicting Biomarker for Delayed Graft Function in Kidney Transplantation. Nephron. 2019;141(4):236-248. doi: 10.1159/000495765. Epub 2019 Jan 11. PMID 30636249